CLINICAL TRIAL: NCT02236351
Title: New Pediatric Patching Method to Improve Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Irene Tintin Tung, Assistant Professor, TCH Ophthalmology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-34627
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Amblyopia; Strabismus
Keywords: patching; pediatric ophthalmology
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Control (Placebo Comparator): Patients assigned to the Control Arm will be taught to apply their patches using the standard technique -- applying the patch evenly and flatly around the orbit.
  Interventions: Device: Pinch Patch/ flat Patch
- Pinched Patch (Experimental): Patients assigned to the Pinched Patch Arm will be taught to apply their patches after pinching the middle of the superior and inferior edges of the patch so that the patch is convex and the center is raised above the eye.
  Interventions: Device: Pinch Patch/ flat Patch

INTERVENTIONS:
Device: Pinch Patch/ flat Patch

SUMMARY:
This project will assess whether there is a significant difference in compliance with patching in amblyopic patients whose parents are instructed to pinch the superior and inferior edges of the patch before applying (in order to improve comfort) versus patients whose parents are instructed to place the patch evenly around the orbit.

DETAILED DESCRIPTION:
Patients will present to the pediatric ophthalmology clinic at Texas Children's Hospital. If during the course of their standard care visit it is determined by their pediatric ophthalmologist or optometrist that patching is indicated and that the patient meets eligibility criteria for the study, the eye doctor will explain to the patient's parents the need for patching according to the standard protocol and will then mention to them the study being conducted. If they are interested, an investigator will explain the study, allow patients and parents to ask questions, and will then seek written informed consent. Upon consent, a patient will be assigned an ID code that will be written on their signed consent form. Consenting parents will then be randomized into either the control group (taught to apply the patch using the standard method) or the study group ( taught to apply the patch using our modified technique). The standard technique refers to applying the patch evenly and flatly around the orbit, and the modified technique refers to pinching the middle of the superior and inferior edges of the patch before applying so that the patch is convex and the center is raised above the eye in an attempt to improve patient comfort. All patients will be provided with one box of sample patches. In order to mask parents in both groups, these patches will all have a small incision of 3 millimeters on the lateral edges so that parents will be uncertain if they are assigned to the control or study group. An incision of this size will not significantly alter the function of the patch in any way. Patients will have equal odds of being assigned to either the control or study group using a random number generator. Parents will not be told whether the method they are being taught is the standard or modified method, and their eye doctor will not be told whether or not the parents decided to enroll in the study. After using one full box of patches or after one month, whichever comes first, parents will complete a questionnaire about their compliance with the prescribed patching regimen and any difficulties they may have had in patching their child. We will use the Amblyopia Treatment Index Patching Questionnaire designed by the Pediatric Eye Disease Investigator Group, with the addition of several questions related to patients' comfort while patching. Patients will be instructed to return for standard follow-up care as determined by their eye doctor.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed an eye patch by a pediatric ophthalmologist or optometrist to treat either strabismus, anisometropia, or deprivation amblyopia
* Patients aged from birth up to and including 7 years old

Exclusion Criteria:

* Known skin reaction to patch or bandage adhesive

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Survey Responses | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States